CLINICAL TRIAL: NCT04498234
Title: Comparison Between Ultrasound Guided Erector Spinae Plane Block and Paravertebral Block on Acute and Chronic Postmastectomy Pain
Brief Title: Comparison Between U\S Guided Erector Spinaeblock and Paravertebral Block on Acute and Chronic Post Mastectomy Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Romany Gergis Naeem Gendy, assistant lecturer, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Romany SECI
Record Dates: First submitted 2020-07-19; First posted 2020-08-04 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Comparison Between Ultrasound Guided Erector Spinae Plane Block and Para-vertebral Block on Acute and Chronic Post Mastectomy Pain
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- GROUP(A) (CONTROL GROUP) (Experimental): Patients will receive standard regimen of anesthesia .
  Interventions: Procedure: ultrasound guided erector spinae plane block with bupivacaine 0.25% And ultrasound guided Paraveretebral block with bupivacaine 0.25 %
- Group B (Experimental): Patients will receive 0.25% bupivacaine (20 ml ) into interfascial plane below erector spinae muscle at level of T4.
  Interventions: Procedure: ultrasound guided erector spinae plane block with bupivacaine 0.25% And ultrasound guided Paraveretebral block with bupivacaine 0.25 %
- Group C (Experimental): Patients will receive (0.3 ml /kg ) 0.25% bubivicaine divided equially at each level of T2 , T4 and T6 at thoracic paravertebral space .
  Interventions: Procedure: ultrasound guided erector spinae plane block with bupivacaine 0.25% And ultrasound guided Paraveretebral block with bupivacaine 0.25 %

INTERVENTIONS:
Procedure: ultrasound guided erector spinae plane block with bupivacaine 0.25% And ultrasound guided Paraveretebral block with bupivacaine 0.25 % — One groupvwill receive 0.25% bupivacaine (20 ml ) into interfascial plane below erector spinae muscle at level of T4 and the other group willreceive (0.3 ml /kg ) 0.25% bubivicaine divided equially at each level of T2 , T4 and T6 at thoracic paravertebral space .

SUMMARY:
compare between ultrasound guided erector spinae plane block and ultrasound guided paravertebral block on acute and chronic post mastectomy pain

DETAILED DESCRIPTION:
Management of postoperative analgesia following breast surgery extending beyond a simple lumpectomy can sometimes be a challenge, especially when such surgery is being performed as a day-case procedure. Patients undergoing mastectomy have a very high possibility of developing postsurgical pain syndrome, as high as 20% to 50%.There has been some evidence to suggest regional analgesia techniques reduce the incidence of postsurgical pain in patients undergoing mastectomy. This underlines the importance of performing regional anaesthetic and analgesic techniques for postoperative analgesia following breast surgery.There are many techniques of regional analgesia as thorasic epidural block , paravertebral block , PECS1 block ,PECS2 block , and recently erector spinae plan block.Paravertebral blocks have superseded thoracic epidurals when it comes to choice of a regional anaesthesia technique to provide analgesia for breast surgery.The injection of local anaesthetic solution in the paravertebral space results in a unilateral block, which is sensory, motor, and sympathetic. The uptake of the local anaesthetic solution is enhanced due to the absence of fascial sheaths binding the spinal nerves.TPVB produces ipsilateral somatic and sympathetic nerve blockade due to a direct effect of the local anesthetic on the somatic and sympathetic nerves in the TPVS, extension into the intercostal space laterally, and the epidural space medially. Ultrasound-guided erector spinae plane (US-ESP) block is a novel analgesic technique, in which local anaesthetic is injected into fascial plane deep to erector spinae muscle. It is possible to block the dorsal and ventral rami of the spinal nerve depending on the level of injection and amount of local anaesthetic injected. Erector spinae block (ESP) leads to effective post-operative analgesia where it is performed at T4-5 level for breast cancer and thoracic surgery , when performed bilaterally it has been reported to be as effective as thoracic epidural analgesia.The drug spreads in craniocaudal fashion over several levels as the erector spinae fascia extends from nuchal fascia cranially to the sacrum caudally. Forero et al. recently described US-ESP block for thoracic neuropathic pain. This block could be effective in both acute post-operative thoracic and abdominal surgeries and also neuropathic pain in these regions.

ELIGIBILITY:
Inclusion Criteria:

1. Gender : female .
2. Age : 20 to 70 years old .
3. Scheduled for : either left or right modified radical mastectomy (MRM)
4. Physical status : American society of anesthesiologists (ASA) physical status I and II.

Exclusion Criteria:

1-ASA > III 2 -age> 70 years old. 3-patients refusal to the procedure. 4-Infection of the skin at or near site of needle puncture. 5- Coagulopathy . 6- Drug hypersensitivity or allergy to the studied drugs. 7- Central or peripheral neuropthy . 8-Pre-operative opoid consumption ( within 24 hours preoperative ) 9- Anomalies of the vertebral column .

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
analgesic requirement | 24 hours
  Total morphine consumption during first 24 hours post operatively.

SECONDARY OUTCOMES:
stress response | 24 hours
  Effect on stress response: serum level of cortisol and noradrenaline (immediately preoperative, after intubation, immediately postoperative, and after 24 hours postoperative)
Chronic post mastectomy pain | 6 month
  Chronic post mastectomy will be assessed at pain clinic at 1st, 3rd, 6 th month postoperatively using (LANSS ) score .

CONTACTS AND LOCATIONS:
Overall Officials: Romany G. Naeem, MSc, Principal Investigator — assistant lecturer
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt

REFERENCES:
- [Derived] Amr SA, Othman AH, Ahmed EH, Naeem RG, Kamal SM. Comparison between ultrasound guided erector spinae plane block and paravertebral block on acute and chronic post mastectomy pain after modified radical mastectomy: randomized controlled trial. BMC Anesthesiol. 2024 Nov 21;24(1):420. doi: 10.1186/s12871-024-02810-4. PMID 39574036